CLINICAL TRIAL: NCT00446524
Title: A 54-week Extension to the Multi-center, Randomized, Double-blind, Parallel-group, Placebo-controlled, Factorial Study to Evaluate the Efficacy and Safety of VAA489 (Valsartan and Amlodipine Combined) and Alone in Essential Hypertensive Patients - Long Term Study of VAA489 in Patients With Essential Hypertension (Extension From A1301 Study)
Brief Title: Long Term Study of Valsartan and Amlodipine in Patients With Essential Hypertension (Extension to Study CVAA489A1301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489A1302
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
Keywords: Hypertension, Valsartan, Amlodipine, high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine; Valine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valsartan + Amlodipine 80/5 mg (Experimental): Valsartan 80 mg or Amlodipine 5 mg ---> Valsartan + Amlodipine 80 / 5 mg
  Interventions: Drug: Valsartan + Amlodipine besilate
- Valsartan + Amlodipine 80/5 mg + Diuretic (Experimental): Valsartan + Amlodipine 80 / 5 mg + Diuretic
  Interventions: Drug: Valsartan + Amlodipine besilate

INTERVENTIONS:
Drug: Valsartan + Amlodipine besilate — During the run-in period, either Valsartan 80 mg or Amlodipine 5 mg tablet was given once daily. Throughout the Valsartan + Amlodipine treatment period, a Valsartan + Amlodipine tablet 80/5 mg was given once daily at around 8:00 AM in the morning.
  Other Names: Valsartan, Amlodipine besilate, VAL, AML

SUMMARY:
The purpose of this study is to evaluate long-term safety and tolerability of once daily administration of the combination of Valsartan and Amlodipine 80/5 mg for 52 weeks in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who successfully complete the core study (Study CVAA489A1301.
* Patients whose blood pressure at Visit 7 of the Study CVAA489A1301 had to be well controlled defined as MSDBP < 90 mmHg and MSSBP < 140 mmHg. At the investigator's or sub-investigator's discretion, those patients who were not well controlled (MSDBP ≥ 90 mmHg or MSSBP ≥ 140 mmHg), and whose MSDBP was < 100 mmHg and MSSBP was < 160 mmHg might participate in the extension if this was considered an acceptable level of blood pressure control for the patient.
* Male or female outpatients.
* Patients who have written informed consent to participate in this study.

Exclusion Criteria:

* Presence of major protocol violation in Study CVAA489A1301.
* Patients who experienced any adverse events considered serious and drug related in Study CVAA489A1301.
* Patients who experienced any adverse events considered serious and drug related in Study CVAA489A1301.
* Patients who are considered unlikely to comply with the requirements specified in the protocol by the investigator or sub-investigator.
* Patients who have gout or gouty arthritis.
* Patients hypersensitive to diuretics (except for potassium sparing diuretics).

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety assessed by serious and non-serious adverse events | 12 months
  No new unexpected AE's were observed in long-term treatment with VAA 80/5 mg. There were no deaths during the study. The SAEs were rare, with 9 patients (2.5%) reporting 10 events (1 patient experienced 2 SAEs). These events were not clustered to any particular primary system organ class and only 2 events the investigators could not excluded a relationship to study drug. The events that occurred were expected in this study population and/or were known to be associated with either valsartan or amlodipine. AEs leading to discontinuation occurred in 14 patients (3.8%).

SECONDARY OUTCOMES:
Efficacy assessed by the changes-from baseline measurements in mean sitting diastolic blood pressure, mean sitting systolic blood pressure, standing diastolic blood pressure, and standing systolic blood pressure | 12 months
  Clinically meaningful reductions in MSDBP and MSSBP were observed after 2 weeks of VAA 80/5 mg treatment and were maintained until the end of the 52-week VAA treatment period. The MSDBP and MSSBP were controlled below 85 mmHg and 130 mmHg, respectively for the entire 52-week VAA treatment period. At endpoint the MSDBP was controlled below 80 mmHg.
Laboratory tests | 12 months
  Laboratory changes observed with the long-term administration of VAA 80/5 mg were consistent with the known effects of each monotherapy agent.
Vital signs | 12 months
  Mean changes from baseline at endpoint were small and clinically unremarkable in extension population for weight, sitting/standing pulse values.
  AEs related to abnormal vital signs were rare during the VAA treatment period. No patient reported orthostatic hypotension as an AE. Only one patient (PID 0045/00007) was discontinued from the study due to blood pressure decreased and dizziness.
Electrocardiogram (ECG) | 12 months
  None of the patients reported shifting from clinically non-significant to clinically significant ECG abnormality. However, three patients experienced clinically significant ECG abnormalities and were reported as AEs during the VAA treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Novartis Investigative Site, Fukuoka, Japan